CLINICAL TRIAL: NCT06933706
Title: Losartan to Improve Outcomes After Multi-ligament Knee Injury
Acronym: LION
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: University of Kentucky (Other); Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Cale Andrew Jacobs, PhD, Assistant Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025P000672
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Multi-ligament Knee Injury
Keywords: knee dislocation; multi-ligament knee injury; losartan
MeSH Terms: conditions — Knee Dislocation | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Losartan (Experimental): Participants randomized to the Losartan arm will be asked to take 25 mg of losartan per day for 30 days.
  Interventions: Drug: losartan 25 mg
- Placebo (Placebo Comparator): Participants randomized to the Placebo arm will be asked to take one placebo capsule per day for 30 days.
  Interventions: Other: Placebo capsule

INTERVENTIONS:
Drug: losartan 25 mg — Losartan is an angiotensin-II inhibitor that modulates the renin-angiotensin system by blocking the activation of angiotensin type 1 receptors, thus preventing binding with angiotensin-II and decreasing blood pressure. Losartan has a broader therapeutic potential for muscle healing and treatment for diseases ranging from rheumatoid arthritis, osteoarthritis, chronic kidney disease, Marfan syndrome, and fatty liver. TGF-β plays an active role in fibrosis leading to the formation of adhesions and scar tissue. By limiting the formation of adhesions and scar tissue, losartan may reduce pain, myofibroblast activity, synovitis, fibrosis, and cartilage degeneration.
  Arms: Losartan
Other: Placebo capsule — The placebo capsule will look identical to the active study drug, but will not have any active ingredient and will be filled with corn starch
  Arms: Placebo

SUMMARY:
Multi-ligament knee injuries (MLKIs) can occur during military training, sports injuries, or traumatic events such as motor vehicle accidents and can be devastating events. These complex injuries involving disruption of 2 or more ligaments often coincide with injuries to arteries, nerves, tendons, menisci, and/or fractures and can be devastating events. MLKIs often require complex treatments nearly 2 in 5 patients suffer complications after surgery. Loss of knee range of motion is the most common complication and is associated with military separation. There are also long-term effects of motion loss, as the need for motion-restoring surgery after MLKI is associated with an increased risk of osteoarthritis within 5 years of surgery. A person's ability to perform both activities of daily living and higher demand physical activities is often impaired both in the short and long term. In fact, only 1 in 3 people return to high-level sport after MLKI. The purpose of this translational randomized clinical trial is to determine if a 30-day course of oral Losartan improves a person's ability to return to work or sport, range of motion and strength, and reduce knee inflammation in the first year after surgical treatment of an MLKI.

DETAILED DESCRIPTION:
Whether the result of military training, a sports injury, or trauma, multi-ligament knee injuries (MLKIs) can be devastating events. MLKI treatment is complex and 38% of all patients report postoperative complications. Loss of knee range of motion (ROM) is the most common complication and is significantly associated with military separation. There are long-term effects of ROM loss, as the need for motion-restoring surgery after MLKI was a significant predictor of physician-diagnosed osteoarthritis within 5 years of surgery. An individual's ability to perform both activities of daily living and higher demand physical activities is thus frequently impaired both in the short and long term. Losartan, an angiotensin receptor blocker, is an FDA-approved treatment for hypertension but because of its multiple mechanisms of action, this low-cost and widely available medication could be repurposed to improve outcomes after MLKI.

Objectives: The purpose of this study is to determine if a 30-day course of oral losartan will improve a person's ability to return to duty or sport within 12 months post-surgery, improve range of motion and strength, and reduce synovitis and capsular thickening after MLKI.

Specific Aims and Study Design: The LION Trial is a double-blind Randomized Controlled Trial to compare the losartan versus placebo with the primary outcome variable being Cincinnati Occupational Rating Scale scores 12 months after surgery. Ninety patients enrolled and will be randomized to take either 25 mg/day of losartan or oral placebo for the first 30 days after surgery. Assessments will include patient-reported outcomes, time to return to duty/sport, knee ROM, isokinetic strength testing, and quantitative ultrasound assessments of synovitis and capsular thickening. Data will be collected at 4 time points: preoperative, after completing the 30-day course of study medication, and 6 months and 12 months after surgery. The investigators will test the following specific aims:

Aim 1: Determine if a 30-day postoperative course of losartan improves the ability to return to duty or sports and patient-reported outcomes when compared to placebo following MLKI.

Aim 2: Assess whether losartan results in more symmetric knee range of motion and quadriceps strength following MLKI when compared to placebo.

Aim 3: Compare ultrasound measures of capsular thickening and synovitis between groups treated with losartan versus placebo following surgical treatment of MLKI.

ELIGIBILITY:
Inclusion Criteria:

* Multi-ligament knee injury defined as a complete grade III injury of 2 or more ligaments
* At least one ligament surgically reconstructed or repaired
* Willingness to comply with the study protocol and assessments

Exclusion Criteria:

* Allergic to any active or inactive ingredient of losartan
* Pregnant, planning to become pregnant, or sexually active females choosing not to use effective means of contraception during the 30-day course of losartan
* Those at increased risk of losartan related side effects including those with severe renal insufficiency, hepatic disease, hypotension, and/or hyperkalemia
* Have a history of prior knee ligament surgery of the involved knee
* Undergoing staged surgical procedures in the treatment of MLKI
* Have a traumatic brain injury that limits their ability to participate in their postoperative care or any condition that would preclude the ability to comply with postoperative rehabilitation
* Have a concomitant injury or underwent a surgical procedure that will preclude the ability to perform range of motion exercises (i.e. surgery for extensor mechanism rupture or avulsion, vascular graft surgery)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Cincinnati Occupational Rating Scale (CORS) | Baseline, 1 month, 6 months, and 12 months
  The CORS is a valid and reliable 7-item scale that quantifies the hours or number of times a patient performs the following activities: sitting, standing/walking, walking on uneven ground/turning/twisting, climbing, squatting, as well as the frequency of lifting/carrying and the pounds carried. Scores range from 0 to 60 with greater scores being indicative of more strenuous work activities.

SECONDARY OUTCOMES:
Medication Adherence | 1 month
  By counting the number of pills remaining in the participant's medication bottle, we will determine the percentage of the study drug that was taken.
Time to return to work or sport | 6 months, 1 year
  Beginning 6 months after surgery, participants will be contacted biweekly via their self-selected method (phone, text, or email) to determine the date that they returned to their pre-injury level or work and/or sport.
International Knee Documentation Committee Subjective Knee Form (IKDC) | Baseline, 1 month, 6 months, and 12 months
  The IKDC is an 18 item instrument has been shown to be valid, reliable, and responsive, and has been previously used to assess outcomes following MLKI procedures. Scores range from 0 to 100 with 100 higher scores indicative of less pain and better knee function.
Pain Visual Analogue Scale (VAS) | Baseline, 1 month, 6 months, and 12 months
  Participants will be asked to rate their pain on a 10 cm scale in 3 different scenarios: worst pain in the past 24 hours, best pain in the past 24 hours, and average pain in the past 24 hours
Knee Range of Motion | Baseline, 1 month, 6 months, and 12 months
  Bilateral knee flexion and extension range of motion will measured using a long-arm goniometer.
Quadriceps Strength | 6 months, 1 year
  Quadriceps strength will be assessed bilaterally using an isokinetic dynamometer 6 and 12 months after surgery. Peak torque of the operative limb will be expressed as a percentage of the peak torque of the non-operative limb, which is termed the limb symmetry index.
Synovitis Grade | 1 month, 6 months, and 12 months
  Dynamic ultrasound will be used to assess the grade of synovitis. Superb microvascular imaging (SMI) will be used to assess synovitis. SMI is similar to Power Doppler; however, visualizes smaller, slower velocity vessels, and as such, SMI has been found to be more sensitive in the assessment of knee synovitis. Participants will be positioned supine with knees in 30° of flexion. Longitudinal suprapatellar scans will be acquired in 3 standardized regions defined by the midline, lateral, and medial patellar poles. Synovitis will be visually graded by a trained radiologist as none, mild, moderate, or severe based on the percentage of the area of interest with visible SMI signal.

CONTACTS AND LOCATIONS:
Overall Officials: Cale Jacobs, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (3):
- United States (3):
  - University of Kentucky, Lexington, Kentucky
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Mass General Brigham, Foxborough, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
IPD from this project will be made available to the research community and to the public at large. Data will be shared through the Harvard Dataverse data repository. A rich dataset will be created which will include patient demographic information, patient-reported outcomes, isokinetic strength, range of motion, and ultrasound assessments of knee synovitis. Demographic information will include patient age, sex, race, ethnicity, body mass index, injury history, intraoperative findings, and surgical treatment. Patient-reported outcomes will include the Cincinnati Occupational Rating Scale (CORS) scores, International Knee Documentation Committee (IKDC) scores, and VAS pain scores
Time Frame: IPD will be made available after data analysis has been completed and the primary study manuscript has been accepted for publication (anticipated March 2030), and will remain available for a minimum of 7 years (anticipated March 2037).
Access Criteria: The project team will make their data available as widely and as freely as possible while safeguarding the privacy of participants and protecting confidential and proprietary data. Furthermore, any research resources will be shared in line with the policies adopted by DOD for the purposes of this grant. Data will be made publicly available, and requestors will be required to complete a data-sharing agreement with Brigham and Women's Hospital. The purpose of the data-sharing agreement is to ensure data security at the recipient site and clarify that manipulating the data for the purposes of identifying subjects is strictly prohibited. No limits or caveats for co-authorship will be required as a precondition for receiving data.